Clinical Evaluation of a Reusable Multifocal Optical Design in a Presbyopic Population Phase II

Protocol CR-6372

Version: 2.0 Amendment 1

Date: 25 October 2019

Investigational Products: JJV Investigational senofilcon A Multifocal Contact Lens and 1-Day Acuvue® Moist Brand Multifocal Contact Lens

Key Words: Presbyopia, Multifocal, etafilcon A, senofilcon A, Daily Wear, Daily Disposable, Reusable, Dispensing, Randomized

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| TABLE | E OF CONTENTS | |
|---|---|---|
| SPONS | OR NAME AND ADDRESS | 6 |
| MEDIC | AL MONITOR | 6 |
| AUTHO | ORIZED SIGNATURES | 7 |
| CHANG | GE HISTORY | 8 |
| SYNOP | SIS | 9 |
| COMM | ONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | 14 |
| 1. IN | TRODUCTION AND BACKGROUND | 16 |
| 1.1. | Name and Descriptions of Investigational Products | 16 |
| 1.2. | Intended Use of Investigational Products | 16 |
| 1.3. | Summary of Findings from Nonclinical Studies | 16 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 16 |
| 1.5.<br>Study | Relevant Literature References and Prior Clinical Data Relevant to Propos 17 | ed Clinica |
| 2. ST | UDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 18 |
| 2.1. | Objectives | 18 |
| 2.2. | Endpoints | 18 |
| 2.3. | Hypotheses | 19 |
| 3. TA | RGETED STUDY POPULATION | 20 |
| 3.1. | General Characteristics | 20 |
| 3.2. | Inclusion Criteria | 20 |
| 3.3. | Exclusion Criteria. | 20 |
| 3.4. | Enrollment Strategy | 21 |
| 4. ST | UDY DESIGN AND RATIONALE | 21 |
| 4.1. | Description of Study Design | 21 |
| 4.2. | Study Design Rationale | 22 |
| 4.3. | Enrollment Target and Study Duration | 22 |
| 5. TE | ST ARTICLE ALLOCATION AND MASKING | 22 |
| 5.1. | Test Article Allocation | 22 |
| 5.2. | Masking | 22 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 23 |
| 6. ST | UDY INTERVENTION | 23 |
| 6.1. | Identity of Test Articles. | 23 |
| 6.2 | Ancillary Supplies/Products | 24 |

| 6.3. Administration of Test Articles | 24 |
|----------------------------------------------|-------------------------|
| 6.4. Packaging and Labeling | 25 |
| 6.5. Storage Conditions | 25 |
| 6.6. Collection and Storage of Samples | 25 |
| 6.7. Accountability of Test Articles | 25 |
| 7. STUDY EVALUATIONS | 27 |
| 7.1. Time and Event Schedule | 27 |
| 7.2. Detailed Study Procedures | |
| VISIT 1 | |
| VISIT 2 | 39 |
| VISIT 3 | 44 |
| VISIT 4 | 47 |
| VISIT 5 | |
| VISIT 6 | 58 |
| FINAL EVALUATION | 60 |
| 7.3. Unscheduled Visits | 61 |
| 7.4. Laboratory Procedures | |
| 8. SUBJECTS COMPLETION/WITHDRAWA | |
| _ | 63 |
| 8.2. Withdrawal/Discontinuation from the Stu | ıdy 63 |
| 9. PRE-STUDY AND CONCOMITANT INTE | |
| 9.1. Systemic Medications | 64 |
| 10. DEVIATIONS FROM THE PROTOCOL | 65 |
| 11. STUDY TERMINATION | 65 |
| 12. PROCEDURE FOR HANDLING PRODUC | CT QUALITY COMPLAINTS66 |
| 13. ADVERSE EVENTS | 67 |
| 13.1. Definitions and Classifications | 67 |
| 13.2. Assessing Adverse Events | 69 |
| - | 69 |
| 13.2.2. Severity Assessment | 70 |
| - | erse Events70 |
| 13.4. Reporting Adverse Events | 71 |
| 13.4.1. Reporting Adverse Events to Spon | sor |

| | 13.4. | <ol> <li>Reporting Adverse Events to the Responsible IEC/IRB and Health Auth</li> <li>72</li> </ol> | orities |
|---|---|---|---|
| | 13.4. | 3. Event of Special Interest | 72 |
| 13 | 3.5. | Reporting of Pregnancy | 73 |
| 14. | ST | ATISTICAL METHODS | 73 |
| 14 | <b>1</b> .1. | General Considerations | 73 |
| 14 | 1.2. | Sample Size Justification | 73 |
| 14 | 1.3. | Analysis Populations | 74 |
| 14 | 1.4. | Level of Statistical Significance | 75 |
| 14 | 1.5. | Primary Analysis | 75 |
| 14 | 1.6. | Secondary Analysis | 75 |
| 14 | 1.7. | Other Exploratory Analyses | 75 |
| 14 | 1.8. | Interim Analysis | 76 |
| 14 | 1.9. | Procedure for Handling Missing Data and Drop-Outs | 76 |
| 14 | 4.10. | Procedure for Reporting Deviations from Statistical Plan | 76 |
| 15. | DA | ATA HANDLING AND RECORD KEEPING/ARCHIVING | 76 |
| 15 | 5.1. | Electronic Case Report Form/Data Collection | 76 |
| 15 | 5.2. | Subject Record | 77 |
| 15 | 5 1 | 15.3 ClinicalTrials.gov | 77 |
| 16. | DA | ATA MANAGEMENT | 77 |
| 16 | 5.1. | Access to Source Data/Document | 77 |
| 16 | 5.2. | Confidentiality of Information. | 77 |
| 16 | 5.3. | Data Quality Assurance | 78 |
| 17. | CL | INICAL MONITORING | 78 |
| 18. | ET | HICAL AND REGULATORY ASPECTS | 79 |
| 18 | 3.1. | Study-Specific Design Considerations | 79 |
| 18 | 3.2. | Investigator Responsibility | 79 |
| 18 | 3.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 79 |
| 18 | 3.4. | Informed Consent | 80 |
| 18 | 3.5. | Privacy of Personal Data | 81 |
| 19. | ST | UDY RECORD RETENTION | 82 |
| 20. | FI | NANCIAL CONSIDERATIONS | 82 |
| 21. | PU | BLICATION | 83 |
| 22. | RE | FERENCES | 83 |

| APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) 84 |
|---|
| APPENDIX B: PATIENT INSTRUCTION GUIDE (To be provided separately) 116 |
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) |
| APPENDIX D: BINOCULAR OVER REFRACTION |
| APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE |
| APPENDIX F: OCULAR DOMINANCE |
| APPENDIX G: LENS FITTING GUIDE |
| APPENDIX H: |
| LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS |
| EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING 160 |
| DETERMINATION OF NEAR ADDITION |
| NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE 173 |
| LENS FITTING CHARACTERISTICS |
| SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS |
| FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE 185 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS 191 |
| BIOMICROSCOPY SCALE |
| KERATOMETRY PROCEDURE |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION |
| DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE 211 |
| , PATIENT REPORTED OUTCOMES |
| WHITE LIGHT LENS SURFACE WETTABILITY |
| VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE |
| TABLE OF CONTENTS Figure 1: Study Flowchart |
| TABLE OF CONTENTS |
| Table 1: Test Articles 23 Table 2: Ancillary Supplies 22 |
| Table 3: Time and Events |
| Table 4: Disallowed systemic medications (less than 6 months of continual use) |

#### PROTOCOL TITLE, NUMBER, VERSION

Clinical Evaluation of a Reusable Multifocal Optical Design in a Presbyopic Population Phase

II

Protocol Number: CR-6372

Version: 2.0

Date: 25 October 2019

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJV) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR

Name: Thomas R. Karkkainen, OD, MS, FAAO

Title: Sr. Principal Research Optometrist

Address: 7500 Centurion Parkway, Jacksonville, Florida 32256

Email: TKarkkai@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### AUTHORIZED SIGNATURES

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, ICH guidelines, ISO 14155, and the Declaration of Helsinki.

| Author | See Electronic Signature Report Thomas R. Karkkainen, OD, MS, FAAO Sr. Principal Research Optometrist, Clinical Sciences | DATE |
|---|---|---|
| Clinical Operations<br>Manager | See Electronic Signature Report | DATE |
| Biostatistician | See Electronic Signature Report | DATE |
| Data Management | See Electronic Signature Report | DATE |
| Reviewer | See Electronic Signature Report | DATE |
| Approver | See Electronic Signature Report | DATE |

#### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section | Date |
|---|---|---|---|
| | | Number(s) Affected | |
| 1.0 | Tom Karkkainen | Original Protocol | 10-Oct-2019 |
| 2.0 | Tom Karkkainen | -Revised Exclusions #6, #13 and #15 | 25-Oct-2019 |
| | | in the Synopses and Section 3.3 | |
| | | -Grammar and Spelling updated | |
| | | throughout protocol | |
| | | -Figure 1 Flowchart updated | |
| | | -Added Study Instruction to steps | |
| | | 2.18, 2.19, 5.48 and 5.19 | |
| | | -Added further details to masking. | |
| | | -Updated Table 4 in section 9.1 | |
| | | -Version and Date updated throughout | |
| | | protocol | |

#### **SYNOPSIS**

| Clinical Evaluation of a Reusable Multifocal Optical Design |
|---|
| in a Presbyopic Population Phase II IIVC 7500 Centurion Parkway Jacksonville FL 32256 |
| JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Development phase, Phase 2 |
| This study will be registered on ClinicalTrials.gov. |
| Investigational Products: JJV Investigational Multifocal |
| Contact Lens manufactured in senofilcon A material. |
| Approved Products: 1-Day Acuvue® Moist Brand Multifocal |
| Contact Lens. |
| Wear Schedule: The Test and Control lenses are used as |
| daily wear (note: the Test lens will be reusable and the |
| Control lens daily disposable). |
| Replacement Schedule: The Test lens will be replaced at the |
| optimization visit. The Control lens will be replaced after |
| each day of wear as well as the optimization visit. The Test |
| and Control lenses will also be replaced when lost or |
| damaged |
| This primary objective of this pilot study is to evaluate the |
| visual performance of the JJV Investigational senofilcon A |
| Multifocal Contact Lens (Test) made using a new |
| manufacturing process by comparison with 1-Day Acuvue® |
| Moist Brand Multifocal (Control). |
| The accordant chiestive is to evaluate the clinical |
| The secondary objective is to evaluate the clinical |
| performance of the Test lens by comparisons with the control |
| lens in the following areas: |
| • Vision (subjective) |
| • Comfort |
| Slit Lamp Findings |
| <ul> <li>Patients' reported ocular symptoms</li> </ul> |
| Primary Endpoints: |
| Binocular distance, intermediate and near visual performance |
| under different lighting conditions. |
| under different fighting conditions. |
| Secondary Endpoints: |
| Overall quality of vision scores on CLUE scale |
| Overall comfort scores on CLUE scale |
| <ul> <li>Subject reported ocular symptoms</li> </ul> |
| <ul> <li>Slit Lamp Findings</li> </ul> |
| on Lump I manigo |

| Study Design | This is a randomized-controlled, single-masked, crossover clinical trial. There are two study lenses. Each lens will be dispensed for $3 \pm 1$ days and then an optimization visit will occur. The final lens pair will be dispensed for $12 \pm 2$ days and the follow-up on the final lens pair will occur. The second study lenses will then be fit and the above sequence repeated. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). |
|---|---|
| Sample Size | Up to 48 subjects will be enrolled with a target completion of 40 subjects. |
| Study Duration | The study will last approximately 2-4 months. |
| Anticipated Study Population | Healthy male and female volunteers with presbyopia will be invited to participate in the study. Subjects will be adapted soft contact lens wearers in both eyes. Additional information regarding the eligibility of the population can be found in the inclusion/exclusion criteria outlined below. |
| Eligibility Criteria | Potential subjects must satisfy all the following criteria to be enrolled in the study Inclusion Criteria after Screening: 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form. 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol. 3. The subject must be at least 40 years of age and not greater than 70 years of age at the time of consent. 4. Subjects must own a wearable pair of spectacles if required for their distance vision. 5. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration). 6. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire". |

Inclusion Criteria after Baseline:

- 7. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D in each eye.
- 8. The subject's refractive cylinder must be  $\leq$ 0.75 D in each eye.
- 9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
- 10. The subject must have distance best corrected visual acuity of 20/20<sup>-3</sup> or better in each eye.

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria after Screening:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
- 3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
- 5. A history of amblyopia, strabismus or binocular vision abnormality.
- 6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, oral phenothiazines, oral/topical/inhaled anticholinergics, systemic/topical corticosteroids.
- 7. Use of any ocular medication, with the exception of rewetting drops.
- 8. History of herpetic keratitis.
- 9. History of irregular cornea.
- 10. History of pathological dry eye.
- 11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).

| | 13. Any known hypersensitivity or allergic reaction to Optifree®Replenish® multi-purpose care solution, sodium fluorescein or non-preserved rewetting drop solutions. |
|---|---|
| | Exclusion Criteria after Baseline: |
| | <ul> <li>14. Clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.</li> <li>15. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.</li> <li>16. Any current ocular infection or inflammation.</li> <li>17. Any current ocular abnormality that may interfere</li> </ul> |
| D: 11 1 | with contact lens wear. |
| Disallowed Madications/Interpretions | Use of any prescription or over-the-counter (OTC) |
| Medications/Interventions | medications that may affect contact lens wear. |
| | See section 9.1 for details regarding disallowed systemic medications. |
| Measurements and Procedures | See Section 7.2 for the detailed procedures. |
| Microbiology or Other<br>Laboratory Testing | None |
| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any SAE where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss this with the Principal Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study-<br>Specific Materials | Rewetting drops, lens cases, glass vials, saline, Early Treatment Diabetic Retinopathy Study (ETDRS) light cabinet, logMAR charts, and Near logMAR charts. Optifree®Replenish® Multipurpose Disinfecting Contact Solution. |
| Principal Investigator(s) and Study Institution(s)/Site(s) | A full list of Principal Investigators, clinical sites, and institutions is kept separately from the Study Protocol and is included in the study Trial Master File. |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDE Investigational Device Exemption IEC Independent Ethics Committee IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator

PIG Patient Instruction Guide PQC Product Quality Complaint PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Johnson & Johnson Vision (JJV) recently launched a multifocal contact lens, 1-DAY ACUVUE® Moist Multifocal. The lens is the only marketed soft multifocal lens to have its optical design optimized for the changes that occur in pupil size with refractive error. The modality for the lens is daily disposable. There is a desire to evaluate the same optical design in a reusable modality. The purpose of this study is to evaluate a multifocal optical design manufactured from senofilcon A material and compare the visual performance to the 1-DAY ACUVUE® Moist Multifocal.

#### 1.1. Name and Descriptions of Investigational Products

Test Lens: JJV Investigational senofilcon A Multifocal Contact Lens-The lens has the same optical design, diameter, aspheric back surface design as the 1-Day Acuvue<sup>®</sup> Moist Brand Multifocal. The lens is manufactured in senofilcon A.

Control Lens: Marketed 1-Day Acuvue® Moist Brand Multifocal Contact Lenses

#### 1.2. Intended Use of Investigational Products

Both lenses are intended to correct spherical refractive error and presbyopia. The Test lenses are intended to be used as a 2-week, reusable, daily wear lens. The lenses require use of a care system to clean and disinfect the lenses. The control lenses are daily wear lenses that are disposed of at the end of each wear cycle. No care system is required for the control lenses.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding JJV investigational senofilcon A multifocal refer to the latest version of the Investigator Brochure.

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

The Investigational multifocal contact lenses are designed as a continuous asphere providing for the correction of refractive spherical ammetropia and presbyopia. The material is a silicone hydrogel material, senofilcon A.

The 1-Day Acuvue<sup>®</sup> Moist Brand Multifocal Contact Lens is a currently marketed product that is made of the etafilcon-A material. The contact lenses are available as continuous aspheres providing for the correction of a subjects refractive spherical ammetropia and presbyopia.

The intent of the Test lens is daily wear, reusable lens that the subject wears while awake. This lens is not intended for extended wear. Anticipated risks and adverse reactions with this lens are similar to other soft daily wear contact lenses used to correct presbyopia. A listing of examples of adverse reactions is found in the Section 13 of this protocol. The investigator should follow normal clinical guidelines regarding examination and care of subjects who participate in this trial. For the most comprehensive clinical information regarding the JJV Investigational senofilcon A multifocal lens refer to the Investigator Brochure. Additional

details on the 1-Day Acuvue® Moist Brand Multifocal Contact Lens can be found in the package insert in Appendix C.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

JJV has evaluated the test lenses in the previous clinical studies:

A summary of these studies is listed below.

was a dispensing clinical trial with primary end points of logMAR visual acuity at fit and CLUE vision scores at 1 week. The study was a cross-over design with a marketed product serving as the control. There were 32 subjects that completed the study as cohort. The Test lens displayed good visual acuity with the mean distance and intermediate logMAR acuity better than 0.0 and the mean near logMAR acuity better than +0.1 logMAR. This with true of the acuity at the initial fit as well as the 1 week and 2-week visits in the final lens pair. There were two non-ocular adverse events that occurred during the study that were not related to any of the Test lenses.

was a dispensing parallel-ARM study and had a primary endpoint of logMAR visual acuity. There were 149 subjects that completed the study overall with 37 subjects completing in the ARM involving the study lenses that will be used in this study. The lenses displayed clinically acceptable logMAR visual acuity after approximately 2 weeks of wear with the mean bright high contrast binocular logMAR acuity of -0.077, -0.083 and 0.049 for distance, intermediate and near respectively.

had four parallel ARMs with one of the ARMs being the test lenses evaluated in this study along with two other investigational test lenses and a control lens. For the ARM with the lenses tested in this study there were no ocular adverse events reported and one non-ocular that was not related to the test article.

was a dispensing crossover study on myope subjects and had a primary endpoint of subject vision response. There were 53 subjects that completed the study as cohort. The test lenses displayed clinically acceptable logMAR visual acuity after approximately 2 weeks of wear with the mean bright high contrast binocular logMAR acuity of -0.11, -0.07 and 0.06 for distance, intermediate and near respectively. There was one adverse event in the study that was a non-significant temporal conjunctival hyperemia in the right eye after removal of their lenses. The event resolved without any treatment.

was a dispensing crossover study on hyperope subjects and had a primary endpoint of subject vision response. There were 59 subjects that completed the study as cohort. The test lenses displayed clinically acceptable logMAR visual acuity after approximately 2 weeks of wear with the mean bright high contrast binocular logMAR acuity of -0.05, -0.02 and 0.11 for distance, intermediate and near respectively. One subject had a non-ocular serious adverse event of dehydration of moderate severity and received treatment for this event. Although the event was reported as resolved, the subject was permanently discontinued the study. The investigator considered the event to be not related to the study article/study procedure. Three episodes of ocular adverse events were reported. One subject had an ocular AE of non-

significant corneal foreign body of mild severity. The subject did not receive any treatment for this event. The event of non-significant corneal foreign body was reported as resolved and no action was taken with the study article. The investigator considered the event to be not related to the study article/study procedure. A second subject had two episodes (one in each eye) of significant infiltrative event (SIE) of moderate severity. The subject received treatment for these events. Although the events were reported as resolved, the subject was permanently discontinued the study. The investigator considered the events to be related to the study article/study procedure.

was a dispensing crossover study on hyperope subjects and had a primary endpoint of subject vision response. There were 42 subjects that completed the study as cohort. The test lenses displayed clinically acceptable logMAR visual acuity after approximately 2 weeks of wear with the mean bright high contrast binocular logMAR acuity of -0.025, -0.045 and 0.173 for distance, intermediate and near respectively. There was one adverse event in the study that was a non-significant contact lens acute red eye in the right eye. The event was classified as related to the test article and resolved with treatment.

In addition to the above studies, JJV had tested similar optical designs that have been manufactured in a similar material, however those lenses were worn as daily disposable lenses. The lenses were tested in Additional details regarding these studies can be found in the Investigator Brochure.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

This primary objective of this pilot study is to evaluate the visual performance of the JJV Investigational senofilcon A Multifocal Contact Lens (Test) made using a new manufacturing process by comparison with 1-Day Acuvue® Moist Brand Multifocal (Control).

The secondary objective is to evaluate the clinical performance of the Test lens by comparisons with the control lens in the following areas:

- Vision (subjective)
- Comfort
- Slit Lamp Findings
- Patients' reported ocular symptoms

#### 2.2. Endpoints

Primary Endpoint(s)

The primary endpoint is contact lens-corrected visual performance on logMAR scale. This will be evaluated binocularly under high luminance high contrast, Dim luminance high contrast and high luminance low contrast conditions at 4 meters (distance), 64 cm (intermediate) and 40 cm (near) from ETDRS/reduced Guillon-Poling charts at the 2-week follow-up visit. For more details refer to section 7.2 Detailed Study Procedures.

#### Secondary Endpoints:

- Overall quality of vision scores on CLUE scale
- Overall comfort scores on CLUE scale
- Subject reported ocular symptoms
- Slit Lamp Findings

#### Other Endpoints(s)

- Lens fitting characteristics (lens centration, lens movement, overall lens fitting acceptability)
- Average daily wear time (in Hours)
- Corneal staining
- Ocular redness (bulbar and limbal)
- Summary of number of lenses needed to fit (optimize) the subject
- Lens deposits
- Overall handling scores on CLUE scale
- Product performance survey questionnaire

Adverse events, number and reasons for discontinuation, number and reasons for unscheduled. lens replacement including lens damage will be monitored and descriptively evaluated.

CLUE<sup>™</sup> is a validated patient reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE<sup>™</sup> scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120. A 5-point increase in an average CLUE<sup>™</sup> score translates into 10% shift in the distribution of scores for population of soft contact lens wearers.<sup>7</sup>

#### 2.3. Hypotheses

#### Primary Hypotheses:

The Test lens will be non-inferior to the Control lens with respect to binocular contact lens-corrected visual performance at near, intermediate and distance under high luminance high contrast, Dim luminance high contrast and high luminance low contrast conditions. A non-inferiority margin of 0.05 on logMAR scale will be used.

#### Secondary Hypotheses:

No secondary hypotheses will be tested. All secondary endpoints will be evaluated with summary tables (see Section 14 for more details). The following will be calculated:

- Average (SD) comfort scores on CLUE scale by study lens at each follow-up visit
- Proportion of eyes with clinically significant (Grade 3 or 4) slit lamp findings.
- Proportion of eyes with reported ocular symptoms.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Healthy male and female subjects who are habitual soft contact lens wearers will be recruited. Subjects will be at least 40 years of age and not older than 70 years of age. They will be hyperopic and have presbyopia.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

Inclusion Criteria after Screening:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. The subject must be at least 40 years of age and not greater than 70 years of age at the time of consent.
- 4. Subjects must own a wearable pair of spectacles if required for their distance vision.
- 5. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month or more duration).
- 6. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire" (Appendix E).

Inclusion Criteria after Baseline:

- 7. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D in each eye.
- 8. The subject's refractive cylinder must be  $\leq 0.75$  D in each eye.
- 9. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
- 10. The subject must have distance best corrected visual acuity of 20/20<sup>-3</sup> or better in each eye.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria after Screening:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.

- 3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
- 5. A history of amblyopia, strabismus or binocular vision abnormality.
- 6. Use of any of the following medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, oral phenothiazines, oral/topical/inhaled anticholinergics, systemic/topical corticosteroids.
- 7. Use of any ocular medication, with the exception of rewetting drops.
- 8. History of herpetic keratitis.
- 9. History of irregular cornea.
- 10. History of pathological dry eye.
- 11. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
- 12. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 13. Any known hypersensitivity or allergic reaction to Optifree®Replenish® multipurpose care solution, sodium fluorescein or non-preserved rewetting drop solutions.

#### Exclusion Criteria after Baseline:

- 14. Clinically significant (Grade 2 or greater) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 15. Entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions.
- 16. Any current ocular infection or inflammation.
- 17. Any current ocular abnormality that may interfere with contact lens wear.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

The clinical study is a randomized-controlled, single-masked, cross-over clinical trial. There are two study lenses. Each lens will be dispensed for  $3\pm1$  days and an optimization visit will occur. The final lens pair will be dispensed for  $12\pm2$  days and the follow-up on the final lens pair will occur. The second study lenses will then be fit and the above sequence repeated.

#### 4.2. Study Design Rationale

The study is intended to compare two study lens types and the initial performance, in terms of the subjective response after a period of lens dispensing. The lenses are dispensed to determine the subjective responses and the comparison is made after a total of 14-20 days of wear.

The cross-over study design was chosen to control for variables that may impact the lens performance between subjects. A washout period will be used to minimize the chances of a significant carry over effect impacting the primary/secondary endpoints measured in the study.

#### 4.3. Enrollment Target and Study Duration

Up to 48 eligible subjects will be enrolled with 40 targeted to complete the study. The anticipated study duration is approximately 3 months.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral and random fashion using a 2×2 crossover design with 2 lens types and 2 periods. Using a computer-generated randomization scheme provided by the study biostatistician, each subject will randomly be assigned to one of two unique sequences (Test/Control or Control/Test). Randomization will be stratified by site.

Permuted block randomization will be used to avoid bias in the assignment of subjects to treatment, and to enhance the validity of statistical comparisons across treatment groups. Each block will contain two different lens trial sequences.

Randomization must be performed at the initial visit. The following must have occurred prior to randomization:

- Informed consent has been obtained
- It has been determined that the subject meets all the inclusion / exclusion criteria
- Subject history and baseline information has been collected

The order of lens wear will be based on the randomization scheme assigned to the study site. The study site will follow the randomization scheme provided and will complete enrollment according to the randomization list and will not pre-select or assign subjects.

#### 5.2. Masking

This is a single-masked (partial) study with the subjects being masked. Subjects will be aware that there are differences in modalities between lens types however they will not be told anything regarding the optical design other than the design is intended to correct for their spherical refractive error and presbyopia. Subjects will be unaware of the identity of the assigned investigational products. Investigators and clinical site personnel involved in the data collection will be aware of the identity of the assigned investigational products.

The identity of the study lenses will be masked to subjects by over labeling the blister packs with a label containing the study number, lot number, sphere power, add power, expiration date and the randomization codes. Investigators and medical monitor will have access to the decode information translating the randomization codes into Test and Control arms.

Under normal circumstances the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- Investigator or designee (documented on the Delegation Log) will consult the lens
  fitting schedule/randomization scheme to obtain the test article assignment for that
  subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme if applicable
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test Lens | Control Lens |
|---|---|---|
| Name | JJV Investigational Multifocal<br>Contact Lens | 1-Day Acuvue® Moist Brand<br>Multifocal Contact Lens |
| Manufacturer | Johnson & Johnson® Vision, Inc. | Johnson & Johnson® Vision, Inc. |

| Par Charles | | 1 |
|---|---|---|
| Lens Material | senofilcon A | etafilcon A |
| Nominal Base Curve | 8.35 mm | 8.4 mm (labeled) |
| Nominal Diameter (mm) | 14.3 mm | 14.3mm |
| Nominal Distance Powers (D) | +1.00 D to<br>+4.00 D in 0.25 D steps | +1.00 D to +4.00 D in 0.25 D<br>steps |
| Nominal Cylinder Powers (D)<br>and Axes | None | None |
| Nominal ADD Powers (D) | Low, Mid, Hgh | Low, Mid, Hgh |
| Water Content | 38% | 58% |
| Center Thickness | 0.070 mm<br>(-3.00 D) | 0.084 mm<br>(-3.00 D) |
| Oxygen Permeability (Dk) | 122.0 | 28.0 |
| Wear Schedule in Current<br>Study | Daily Wear Reusable | Daily Wear |
| Replacement Frequency | Two Weeks | Daily Disposable |
| Packaging Form (vial, blister, etc.) | Blister | Blister |

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Single-Use Preservative-Free Rewetting Solutions (any of these three options may be supplied) | | |
|---|---|---|---|
| Solution<br>Name/Description | Eye-Cept® Rewetting<br>Drops | ScleralFil® Preservative Free Saline Solution | LacriPure Saline<br>Solution |
| Manufacturer | Optics Laboratory | B&L | Menicon |
| Preservative | Non-Preserved Non-preserved Non-preserved | | |

| | Solution |
|---------------------------|-----------------------------------------|
| Solution Name/Description | OPTI-FREE® Replenish® |
| Solution Name/Description | Multipurpose Disinfecting Solution |
| Manufacturer | Alcon Laboratories |
| Preservative | Myristamidopropyl dimethylamine 0.0005% |
| Pieservanive | polyquaternium-1 0.001% |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subjects meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blisters, as the primary packaging. The test article will be over-labeled to mask the subject to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Event and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits.
- 2. What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

Site Instructions for Test Article Receipt and Test Article Accountability for additional information.

### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1<br>Screening,<br>Baseline,<br>Treatment<br>1 Fitting | Visit 2<br>Treatment 1<br>Follow-up 1<br>Optimization | Visit 3<br>Treatment 1<br>Follow-up 2 | Visit 4 Baseline Treatment 2 Fitting | Visit 5<br>Treatment 2<br>Follow-up 1<br>Optimization | Visit 6<br>Treatment 2<br>Follow-up 2 |
|---|---|---|---|---|---|---|
| Time Point | Day 0 | Day 3±1<br>from V1 | Day 12±2<br>from V2 | Day 7±3<br>from V3<br>Fitting<br>Day 0 | Day 3±1<br>from V4 | Day 12±2<br>from V5 |
| Estimated Visit<br>Duration | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours |
| Statement of<br>Informed Consent | Х | | | | | |
| Demographics | X | , | | | | |
| Medical<br>History/Concomit<br>ant Medications | х | | | | | |
| Adverse Events<br>and Concomitant<br>Medications<br>Review | | x | X | х | x | х |
| Compliance | | X | X | | X | X |

CR-6372, v 2.0


| Visit Information Time Point | Visit 1<br>Screening,<br>Baseline,<br>Treatment<br>1 Fitting<br>Day 0 | Visit 2 Treatment 1 Follow-up 1 Optimization Day 3±1 from V1 | Visit 3 Treatment 1 Follow-up 2 Day 12±2 from V2 | Visit 4 Baseline Treatment 2 Fitting Day 7±3 from V3 | Visit 5 Treatment 2 Follow-up 1 Optimization Day 3±1 from V4 | Visit 6<br>Treatment 2<br>Follow-up 2<br>Day 12±2<br>from V5 |
|---|---|---|---|---|---|---|
| | | | | Fitting<br>Day 0 | | |
| Estimated Visit<br>Duration | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours |
| Habitual Contact<br>Lens Information | X | | | | | |
| Contact Lens<br>History | х | | | | | |
| Wear Time and<br>Comfortable<br>Wear Time with<br>Habitual Lenses | х | | | | | |
| Wear Time and<br>Comfortable<br>Wear Time with<br>Study Lenses | | X | х | | х | х |
| Screening<br>Inclusion/Exclusi<br>on Criteria | х | | | | | |
| Subject Reported<br>Ocular Symptoms | X | Х | х | X | X | х |
| Baseline<br>Questionnaire | X | | _ | | | |

CR-6372, v 2.0



| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 |
|---|---|---|---|---|---|---|
| v isit information | Screening, | Treatment 1 | Treatment 1 | Baseline | Treatment 2 | Treatment 2 |
| | Baseline, | Follow-up 1 | Follow-up 2 | Treatment | Follow-up 1 | Follow-up 2 |
| | Treatment | Optimization | renew up 2 | 2 Fitting | Optimization | ronow up 2 |
| | 1 Fitting | · | | | P | |
| Time Point | Day 0 | Day 3±1 | Day 12±2 | Day 7±3 | Day 3±1 | Day 12±2 |
| | | from V1 | from V2 | from V3 | from V4 | from V5 |
| | | | | Fitting | | |
| | | | | Day 0 | | |
| Estimated Visit | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours |
| Duration | | | | | | |
| CLDEQ-8 | X | | x | | | x |
| Questionnaire | A | | Α | | | Λ |
| Distance and | | | | | | |
| Near Entrance | X | X | X | X | X | X |
| Visual Acuity | | | | 41.0 | | |
| Lens Removal | X | X | X | x (if applicable) | X | X |
| Keratometry | X | | | | | |
| Subjective | | | | | | |
| Refraction and | X | | | | | |
| Distance Visual | Α | | | | | |
| Acuity | | | | | | |
| Near ADD | X | | | | | |
| Determination | Α. | | | | | |
| Ocular | X | | | | | |
| Dominance | | | | | | |
| ADD Refinement | X | | | | | |
| Near Visual | X | | | | | |
| Acuity | 21 | | | | | |
| Biomicroscopy | X | X | X | X | X | X |

CR-6372, v 2.0




| Visit Information Time Point | Visit 1<br>Screening,<br>Baseline,<br>Treatment<br>1 Fitting<br>Day 0 | Visit 2<br>Treatment 1<br>Follow-up 1<br>Optimization | Visit 3<br>Treatment 1<br>Follow-up 2 | Visit 4 Baseline Treatment 2 Fitting Day 7±3 | Visit 5 Treatment 2 Follow-up 1 Optimization Day 3±1 | Visit 6<br>Treatment 2<br>Follow-up 2 |
|---|---|---|---|---|---|---|
| | | from V1 | from V2 | from V3<br>Fitting<br>Day 0 | from V4 | from V5 |
| Estimated Visit<br>Duration | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours |
| Baseline<br>Inclusion/Exclusi<br>on Criteria | Х | | | | | |
| Continuance | | | | X | | |
| Lens Selection | X | x (if modified) | | X | x (if modified) | |
| Lens Insertion | X | X | X | X | X | X |
| 10 Minute<br>Settling | x | x (if modified) | | х | x (if modified) | |
| Visual Satisfaction / Subjective Acceptance | X | х | X | x | x | х |
| Study Lens<br>Distance and<br>Near Visual<br>Acuity | х | x | x | х | х | х |
| Distance Over<br>Refraction and<br>Visual Acuity | X | х | | X | x | |

CR-6372, v 2.0



| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 |
|---|---|---|---|---|---|---|
| v isit information | The second second | The second secon | The state of the s | V 1811 4 Baseline | Treatment 2 | The state of the s |
| | Screening, | Treatment 1 | Treatment 1 | | | Treatment 2 |
| | Baseline, | Follow-up 1 | Follow-up 2 | Treatment | Follow-up 1 | Follow-up 2 |
| | Treatment | Optimization | | 2 Fitting | Optimization | |
| T. D : 1 | 1 Fitting | D 211 | D 1010 | D 512 | D 211 | D 1010 |
| Time Point | Day 0 | Day 3±1 | Day 12±2 | Day 7±3 | Day 3±1 | Day 12±2 |
| | | from V1 | from V2 | from V3 | from V4 | from V5 |
| | | | | Fitting | | |
| | | | | Day 0 | | |
| Estimated Visit | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours |
| Duration | | | | | | |
| Lens Fit | 1000 | | • | • | - | ** |
| Assessment | X | X | X | X | X | X |
| Binocular Over | | | ** | | , | v |
| Refraction | | | X | | | X |
| Lens Deposits | | 2 | X | | | X |
| Lens Wettability | | | X | | | X |
| Visual | | | • | | | ** |
| Performance | | | X | | | X |
| Modifications | X | X | | X | X | |
| Post-Fit PRO | | | | | 12. | |
| Questionnaire | X | X | | X | X | |
| Worn Lens | | •• | | | • | ** |
| Collection | | X | X | | X | X |
| Baseline PRO | х | | | | 5 | |
| Questionnaire | A | | | | | |
| Study Lens PRO | | v | v | | v | v |
| Questionnaire | | X | X | | X | X |
| Distance and | | | | | | |
| Near Exit Visual | X | X | X | X | X | |
| Acuity | 212 | | 100 | | | |

CR-6372, v 2.0




| Visit Information | Visit 1 Screening, Baseline, Treatment 1 Fitting | Visit 2<br>Treatment 1<br>Follow-up 1<br>Optimization | Visit 3<br>Treatment 1<br>Follow-up 2 | Visit 4 Baseline Treatment 2 Fitting | Visit 5<br>Treatment 2<br>Follow-up 1<br>Optimization | Visit 6<br>Treatment 2<br>Follow-up 2 |
|---|---|---|---|---|---|---|
| Time Point | Day 0 | Day 3±1<br>from V1 | Day 12±2<br>from V2 | Day 7±3<br>from V3<br>Fitting<br>Day 0 | Day 3±1<br>from V4 | Day 12±2<br>from V5 |
| Estimated Visit<br>Duration | 2.5 hours | 1.0 hours | 1.5 hours | 2.5 hours | 1.0 hours | 1.5 hours |
| Dispensing<br>Criteria | x | X | | x | x | |
| Instructions | X | X | X | X | X | |
| Schedule Follow-<br>up | X | X | Х | Х | Х | |
| Final Evaluation | | | | | | X |

### 7.2. Detailed Study Procedures

#### VISIT 1

Subjects must report to the visit wearing their habitual contact lenses to accurately assess baseline PRO (CLUE and MRD) performance. If the subject is not wearing their lenses they must be rescheduled.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's age, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |
| 1.5 | Contact Lens History | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). |
| 1.6 | Wear time and<br>Comfortable Wear<br>time with Habitual<br>lenses | Record the subjects wear time and comfortable wear time with their habitual contact lenses. |
| 1.7 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |

| | Visit 1: Baseline | |
|---|---|---|
| Step | Procedure | Details |
| 1.8 | Baseline PRO<br>(CLUE and MRD)<br>and CLDEQ-8<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of their habitual lenses using the PRO questions. |

| 1.9 | Ocular Symptoms | Subjects will respond to a verbal open-ended | |
|---|---|---|---|
| 1.10 | Entrance Visual<br>Acuity | symptoms questionnaire. Distance and near Snellen visual acuity will be measured for each eye with the subject's habitual contact lenses in place. | |
| | | For near measures use the ETDRS 2000<br>Series Chart 1 or 2.<br>The acuity will be recorded to the nearest<br>letter OD, OS and OU. | |
| 1.11 | Lens Removal | Have the subject remove their habitual lenses and store in an approved storage solution. | |
| 1.12 | Keratometry | Keratometry will be performed OD and OS and the steep and flat dioptric power and corresponding meridians recorded. | |
| 1.13 | Subjective<br>Refraction and<br>Distance Visual<br>Acuity | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity to the nearest letter. | |
| | | Note: Best distance visual acuity with sphero-cylindrical refraction must be at least $20/20^{-3}$ in each eye for the subject to be eligible in the study. | |
| 1.14 | Near ADD<br>Determination | The near reading addition will be determined using the binocular crossed cylinder technique (BCC) at 40 cm followed by optimization in a trial frame in step 1.16 below. | |
| 1.15 | Ocular Dominance | Determine the distance ocular dominance with the best distance correction in place using a +1.00-blur test. If the results are equivocal use the sighting dominance test to determine the dominant eye used for the study. | Appendix<br>F |
| 1.16 | ADD Refinement | Place the BCC result in the trial frame and refine the near prescription with trial lenses (or flippers) under binocular conditions. | |
| 1.17 | Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm. Record the near visual acuity OD, OS and OU at 40 cm. | |
| 1.18 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. | |

| | | For the conjunctival redness unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. If any of these slit lamp findings are Grade 2 or higher, the subject will be discontinued. If discontinued a final examination must be completed. |
|---|---|---|
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 1.19 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If so, proceed to lens fitting. If not, complete the final evaluation and discharge the subject. |

| | Visit 1: Treatment 1 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.20 | Randomization and<br>Lens Wear Schedule | Record the randomization ID and lens wear schedule (daily disposable, daily reusable wear). | |
| 1.21 | Lens Selection | Select the lens pair and power based on the Randomization and fitting guide for each eye. Record the test lens parameters (power and lot number). | Appendix<br>G (Fitting<br>Guide) |
| 1.22 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. Complete the Quality Product Complaint form. | |
| 1.23 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. | |
| 1.24 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to | |

| | | read a book, magazine or similar for near | |
|---|---|---|---|
| | | Vision. | |
| 1.25 | Study Lens Distance<br>and Near Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. Note: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity | |
| 1.26 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 1.27 | Lens Fit Assessment | <ul> <li>Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test).</li> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form.</li> </ul> | |
| 1.28 | Modifications | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity OU with the lenses then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or | Appendix<br>G (Fitting<br>Guide) |
| 1.29 | Post-Fit PRO (MRD)<br>Questionnaire | over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 1.21-1.27 will be repeated for each modification. The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms | |
|---|---|---|--|
| | | of the study lenses using the PRO questionnaire. | |
| 1.30 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Note: The distance visual acuity must be at least 20/30 OU for the lenses to be | |
| 1.31 | Dispensing Criteria | <ul> <li>dispensed.</li> <li>The lenses will be dispensed for 2-4 days.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> | |
| 1.32 | Patient Instructions<br>for Daily Disposable<br>Lenses (if<br>applicable) | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required</li> </ul> | |

| | | <ul> <li>number of days until their follow-up visit.</li> <li>No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all</li> </ul> |
|---|---|---|
| | | <ul> <li>unworn study lenses.</li> <li>No cleaning or disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their</li> </ul> |
| | | glasses when not wearing the study lenses. • A patient instruction booklet will be provided. Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor. |
| 1.33 | Patient Instructions for Daily Reusable Wear Lenses (if applicable) | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>OPTI-FREE® Replenish® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> </ul> |

| | | <ul> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> <li>Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor.</li> </ul> |
|---|---|---|
| 1.34 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 3±1 days. Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

#### VISIT 2

The subjects must present to Visit 2 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 2: Treatment 1 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 2.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 2.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 2.3 | Compliance | Record the subject's compliance with wearing the study lenses. |

| | T | | 1 |
|---|---|---|---|
| | | Note: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. | |
| 2.4 | PRO (CLUE)<br>Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. | |
| 2.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 2.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. | |
| 2.7 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU to the nearest letter. Record the results. | |
| | | For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 2.8 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results and distance visual acuity OD and OS. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 2.9 | Determination of Lens Optimization | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity OU with the lenses then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an | Appendix G<br>(Fitting<br>Guide) |

| <u> </u> | | |
|---|---|---|
| 2.10 | Lens Fit Assessment | acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide and steps 1.21-1.27 in Visit 1 Fitting allowing for at least 10 minutes of settling time between each lens modification. Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). • The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear comea) in any gaze • presence of edge lift |
| | | <ul> <li>presence of edge IIIT</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>If either lens is deemed unacceptable, the subject will be discontinued from the study.</li> </ul> |
| | | Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| 2.11 | Collection of<br>unworn lenses (if<br>applicable) | Collect unworn lenses returned by the subject when lens power has been optimized Note: If lens power was not changed allow the subject to use the unworn lenses dispensed at Visit 1 and dispense enough lenses of the same power to last the subject until their next visit. |
| 2.12 | Lens Removal | The study lenses will be removed and discarded. |
| 2.13 | Biomicroscopy | Perform Biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. For the conjunctival redness unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. |

| 2.14 | Insertion of Study | If any of these slit lamp findings are Grade 3 or higher, an AE must be recorded. All AEs must be followed to resolution. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. Dispense the subject a new pair of lenses that |
|---|---|---|
| | Lenses | match the distance and ADD power of the lenses that were removed in Step 2.12 above. |
| 2.15 | PRO (MRD)<br>Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. |
| 2.16 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Note: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
| 2.17 | Dispensing Criteria | <ul> <li>The lenses will be dispensed for 10-14 days.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 2.18 | Patient Instructions for Daily Disposable Lenses | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> </ul> |

| | | A navy long will be approad and warm each |
|---|---|---|
| | | A new lens will be opened and worn each day. |
| | | day. |
| | | Instruct the subject to bring back all |
| | | unworn study lenses. |
| | | No cleaning or disinfecting solutions will |
| | | be used. If determined necessary by the |
| | | Investigator sterile non-preserved |
| | | rewetting drops may be dispensed to be |
| | | used as needed for dryness. |
| | | Subjects will be instructed to wear lenses |
| | | for a minimum of 6 hours a day, every |
| | | day during the study. |
| | | Subjects will be instructed to wear their |
| | | glasses when not wearing the study |
| | | lenses. |
| | | Subjects will be instructed to bring their |
| | | habitual contacts or spectacles to the next |
| | | visit. |
| | | Note: In the event a lens is lost or damaged, |
| | | the subject will return to the investigator site |
| | | for replacement. As much as reasonably possible, a damaged lens should be returned |
| | | to the investigational site and then returned to |
| | | the Sponsor. If lens damage is present, |
| | | complete the Product Quality Complaint |
| | | Form. The lens will be stored in labeled vial |
| | | with sterile saline, and returned to the |
| 2.10 | D. C. A. T. A. C. | Sponsor. |
| 2.19 | Patient Instructions | Instruct the Subject the following: |
| | for Daily Reusable<br>Wear Lenses | The lenses will be worn on a daily wear basis. |
| | vicai Lenses | basis. |
| | | OPTI-FREE® Replenish® solution will be |
| | | used in a rub regime to disinfect and store |
| | | the lenses each night in the lens case provided. |
| | | TC 1 / 1 / 1 |
| | | Investigator sterile non-preserved |
| | | rewetting drops may be dispensed to be |
| | | used as needed for dryness. |

| | | <ul> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their habitual contacts or spectacles to the next visit.</li> </ul> |
|---|---|---|
| | | Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor. |
| 2.20 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 12±2 days. Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

#### VISIT 3

The subjects must present to Visit 3 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 3: Treatment 1 Follow-up 2 | |
|---|---|---|
| Step | Procedure | Details |
| 3.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 3.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |

| 2.2 | C 1: | D 14 1 4 1 4 1 4 | 9 2 |
|---|---|---|---|
| 3.3 | Compliance | Record the subject's compliance with | |
| | | wearing the study lenses. | |
| | | Note: Subjects must have worn lenses for at | |
| | | least 6 hours per day | |
| | | To be counted as a day of wear at this visit | |
| | | the Subject must have worn the study lenses | |
| 4 | | for 6 hours prior to the visit. | |
| 3.4 | PRO (CLUE and | The subject will evaluate the vision | |
| | MRD) and CLDEQ- | characteristics, comfort characteristics, | |
| | 8 Questionnaires | handling characteristics, and visual | |
| | NAME OF TAXABLE PARTY O | symptoms of the study lenses using the PRO | |
| | | questionnaire. | |
| 3.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended | |
| | | symptoms questionnaire | 225 |
| 3.6 | Subjective | Record whether the subject's distance and | 7. |
| | Acceptance | near vision with the lenses is acceptable. | |
| 3.7 | Distance and Near | Measure the distance and near visual acuity | |
| 640,000 | Entrance Visual | OD, OS and OU to the nearest letter. Record | 200 |
| | Acuity | the results. | |
| | 120 | 122 202 32 32 | |
| | | For near measures use the ETDRS 2000 | |
| | | Series Chart 1 or 2. | |
| | | The acuity will be recorded to the nearest | |
| | | letter OD, OS and OU. | |
| 3.8 | Visual Performance | Visual performance will be recorded OD, OS, | <u> </u> |
| 3.0 | Distance (4M) | and OU for the following: | |
| | Intermediate (64 cm) | tale of for the renewing. | |
| | Near (40 cm) | Distance, Bright Illuminance | |
| | real (40 cm) | High and Low Contrast ETDRS Charts | |
| | | 4M- HC#1, HC#2, HC#3 and LC#1, LC#2, | |
| | | LC#3 | |
| | | Near, Bright Illuminance | |
| | | Reduced Guillon-Poling Charts | |
| | | Intermediate (64 cm) High Contrast and Low | |
| | | Contrast | |
| | | Near (40 cm) High Contrast and Low | |
| | | Contrast | |
| | | Series School Wiley White to be a little to be a pro- | |
| | | Distance, Dim Illuminance (with <u>Distance</u> | |
| | | goggles) | |
| | | High Contrast ETDRS Charts | |
| | | 4M-HC#4, HC#5, HC#6 | |
| | | Near, Dim Illuminance (with <u>Near goggles</u> ) | |
| | | Reduced Guillon-Poling charts | |
| | | High Contrast Intermediate (64 cm) and Near | |

| | | (40 cm). | |
|---|---|---|---|
| | | Note: • The room illuminance must be between 7.3 and 7.9 EV (394-597 lux). • Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m2). • Guillon-Poling, Near Chart Luminance Acceptable Range 10.8-11.1 EV (223-274 cd/m2). • Do not use the Mesopic filter for Dim luminance (Dim luminance will be simulated by using the goggles) | |
| 3.9 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix D |
| 3.10 | Lens Fit Assessment | <ul> <li>Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test).</li> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form.</li> </ul> | |
| 3.11 | Lens Deposits | Grade and record the amount of front and back surface lens deposits for both eyes. | |
| 3.12 | Lens Wettability | Grade the wettability of the lenses. | |
| 3.13 | Collection of unworn lenses (if applicable) | Collect unworn lenses returned by the subject. | |

| T D 1 | TT 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |
|---|---|---|
| Lens Removal | 3 | |
| | store in saline in a labeled glass vial. | |
| Biomicroscopy | | |
| | grade the findings. | |
| | For the conjunctival redness 0.5 | - |
| | unit increments will be used in the grading. | |
| | Corneal Staining Assessment | |
| | will be graded in 1.0 increments. | |
| | If any of these slit lamp findings are Grade 3 | |
| | or higher, an AE must be recorded. All AEs | |
| | must be followed to resolution. | |
| | If the clearance of the fluorescein needs to be | |
| | expedited, preservative-free rewetting drops | |
| | may be instilled. | |
| Distance and Near | Distance and near Snellen visual acuity will | |
| Exit Visual Acuity | be measured for each eye with the subject's | |
| Annual record and a second record and a second seco | | |
| | For near measures use the ETDRS 2000 | |
| | Series Chart 1 or 2. | |
| | The acuity will be recorded to the nearest | |
| | letter OD, OS and OU. | |
| Schedule | The subject will complete a wash-out period | |
| Follow-up | and be scheduled to return for their next visit | |
| • | in 7±3 days. | |
| | 1 | |
| | NOTE: Subject may wear their habitual | |
| | washout period. | |
| | Exit Visual Acuity Schedule | store in saline in a labeled glass vial. NOTE: Lenses do not need to be stored in a refrigerator. Perform Biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. For the conjunctival redness O.5 unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. If any of these slit lamp findings are Grade 3 or higher, an AE must be recorded. All AEs must be followed to resolution. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. Distance and Near Exit Visual Acuity Distance and near Snellen visual acuity will be measured for each eye with the subject's habitual correction in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Schedule Follow-up The subject will complete a wash-out period and be scheduled to return for their next visit in 7±3 days. NOTE: Subject may wear their habitual spectacles or contact lenses during the |

### VISIT 4

The subjects may present to Visit 4 wearing their habitual spectacles or contact lenses, if required for their distance vision.

| | Visit 4: Baseline Treatment 2 | |
|---|---|---|
| Step | Procedure | Details |
| 4.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. |

| | 1 | Telefon on the telefon of telefon of the telefon of t | |
|---|---|---|---|
| | | Record any adverse events or medical history | |
| | | changes from the previous study visit. | |
| 4.2 | Subject Reported | Subjects will respond to a verbal open-ended | V2 - 3 |
| | Ocular Symptoms | symptoms questionnaire. | no. |
| 4.3 | Distance and Near | Distance and near Snellen visual acuity will | |
| | Entrance Visual | be measured for each eye with the subject's | 11.5 |
| | Acuity | habitual correction in place. | |
| | 200 | | |
| | | For near measures use the ETDRS 2000 | |
| | | Series Chart 1 or 2. | |
| | | The acuity will be recorded to the nearest | |
| | | letter OD, OS and OU. | |
| 4.4 | Lens Removal (if | Have the subject remove their habitual lenses | |
| | applicable) | and store in an approved storage solution. | us s |
| 4.5 | Biomicroscopy | FDA Slit Lamp Classification Scale will be | |
| | 507(50) | used to grade the findings and determine | |
| | | eligibility. | |
| | | For the conjunctival redness 0.5 | |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment | |
| | | will be graded in 1.0 increments. | |
| | | If any of these slit lamp findings are Grade 3 | |
| | | or higher, an AE must be recorded. All AEs | |
| | | must be followed to resolution. After | |
| | | resolution the subject will be discontinued | |
| | | and Final evaluation completed | |
| | | r | |
| | | If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free rewetting drops | |
| | | may be instilled. | |
| 4.6 | Continuance | Determine whether the subject is eligible to | |
| | | continue in the study based on the | |
| | | examination findings. | |

| | | Visit 4: Treatment 2 Lens Fitting | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.7 | Lens Wear Schedule | Record the lens wear schedule (daily disposable, daily reusable wear). | 20-2- AN |
| 4.8 | Lens Selection | Select the lens pair and power based on the Randomization and fitting guide for each eye. Record the Test lens parameters (power and lot number). | Appendix<br>G (Fitting<br>Guide) |

| 4.9 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. |
|---|---|---|
| | | Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. Complete the Quality Product Complaint form. |
| 4.10 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. |
| 4.11 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. |
| 4.12 | Study Lens Distance<br>and Near Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 4.13 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |
| 4.14 | Lens Fit Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Iimbal exposure at primary gaze or with extreme eye movement; edge lift; excessive movement in primary and up gaze; or |

| | | • insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up. If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |
|---|---|---|---|
| 4.15 | Modifications | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual acuity OU with the lenses then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 4.8-4.14 will be repeated for each modification | Appendix<br>G (Fitting<br>Guide) |
| 4.16 | Post-Fit PRO (MRD) Questionnaire Distance and Near | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. Distance and near Snellen visual acuity will | |
| 4.18 | Exit Visual Acuity Dispensing Criteria | be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Note: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. The lenses will be dispensed for 2-4 days. | |

| | | Distance Snellen acuity equal to or<br>better than 20/30 OU |
|---|---|---|
| | | Subject must indicate that the vision is acceptable. |
| | | Subject must indicate that the comfort of the lenses is acceptable. |
| | | Lenses must have an acceptable general lens fit. |
| 4.19 | Patient Instructions for Daily Disposable Lenses (if applicable) | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>No cleaning or disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial</li> </ul> |
| | | with sterile saline, and returned to the Sponsor. |

| 4.20 | Patient Instructions for Daily Reusable Wear Lenses (if applicable) | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>OPTI-FREE® Replenish® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> <li>Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial</li> </ul> |
|---|---|---|
| | | with sterile saline, and returned to the Sponsor. |
| 4.21 | Schedule | The subject will be scheduled to return for |
| | Follow-up | their follow-up appointment in 3±1 days. |
| | | Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

#### VISIT 5

The subjects must present to Visit 5 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 5: Treatment 2 Follow-up 1 | |
|------|----------------------------------|---------|
| Step | Procedure | Details |

| 5.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
|---|---|---|
| 5.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 5.3 | Compliance | Record the subject's compliance with wearing the study lenses. Note: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 5.4 | PRO (CLUE) Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. |
| 5.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 5.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 5.7 | Distance and Near<br>Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. |
| | | For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 5.8 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results and distance visual acuity OD and OS. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |

| 7.0 | D | If the online the new arts are satisficated as well as | 1: 0 |
|---|---|---|---|
| 5.9 | Determination of | If the subject reports unsatisfactory vision, or is unable to obtain 20/30 distance visual | Appendix G |
| | Lens Optimization | acuity OU with the lenses then a modification | (Fitting<br>Guide) |
| | | must be attempted. | Guide) |
| | | If the subject reports satisfactory vision with | |
| | | the lenses a modification is not required, | |
| | | however at the Investigator's discretion and | |
| | | based upon their findings on the measured | |
| | | visual acuity and/or over- refraction the | |
| | | investigator may make a modification. | |
| | | Up to two attempts at modification are | |
| | | permitted if necessary, in order to achieve an | |
| | | acceptable distance and near binocular | |
| | | performance for the subject, and to enable | |
| | | them to wear that particular lens type. | |
| | | Follow the fitting guide and steps 4.8-4.14 in | |
| | | Visit 4 Fitting, allowing for at least 10 minutes of settling time between each lens | |
| | | modification. | |
| 5.10 | Lens Fit Assessment | Evaluate and grade lens centration, primary | |
| 0.10 | | gaze movement, upgaze movement and | |
| | | tightness (push-up test). | |
| | | The subject should not proceed to wear the | |
| | | lenses if any of the following is observed: | |
| | | • presence of limbal exposure (appearance | |
| | | of clear cornea) in any gaze | |
| | | presence of edge lift | |
| | | presence of unacceptable movement | |
| | | (excessive or insufficient) in <u>all three</u> | |
| | | movement categories (primary gaze, | |
| | | upgaze, and push-up). | |
| | | If oith on long is downed were a served to | |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. | |
| | | Remove the lenses, perform a slit-lamp | |
| | | evaluation, and complete the Final | |
| | | Evaluation form. | |
| 5.11 | Collection of | Collect unworn lenses returned by the subject | |
| | unworn lenses (if | when lens power has been optimized | |
| | applicable) | | |
| | | <b>Note:</b> If lens power was not changed allow | |
| | | the subject to use the unworn lenses | |
| | | dispensed at Visit 4 and dispense enough | |

| | | 1 | is . |
|---|---|---|---|
| | | lenses of the same power to last the subject until their next visit. | |
| 5 12 | Lens Removal | PORTO ACCOUNT OF THE PORTO ACC | |
| 5.12 | Lens Removal | The study lenses will be removed and discarded. | |
| 5.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. For the conjunctival redness unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. If any of these slit lamp findings are Grade 3 or higher, an AE must be recorded. All AEs must be followed to resolution. | |
| 000 - 100 TOO | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. | |
| 5.14 | Insertion of Study<br>Lenses | Dispense the subject new lenses that match<br>the distance and ADD power of the lenses<br>that were removed in Step 5.12 above. | |
| 5.15 | PRO (MRD)<br>Questionnaire | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. | , |
| 5.16 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. Note: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. | |
| 5.17 | Dispensing Criteria | <ul> <li>The lenses will be dispensed for 10-14 days.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> </ul> | |

| | | · |
|---|---|---|
| | | • Lenses must have an acceptable general |
| | | lens fit. |
| 5.18 | Patient Instructions for Daily Disposable Lenses | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>No cleaning or disinfecting solutions will be used. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their habitual contacts or spectacles to the next</li> </ul> |
| 5.19 | Patient Instructions for Daily Reusable Wear Lenses | Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor. Instruct the Subject the following: The lenses will be worn on a daily wear basis. |

| | | <ul> <li>OPTI-FREE® Replenish® solution will be used in a rub regime to disinfect and store the lenses each night in the lens case provided.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their habitual contacts or spectacles to the next visit.</li> </ul> |
|---|---|---|
| | | Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline, and returned to the Sponsor. |
| 5.20 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 12±2 days. Note: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

### VISIT 6

The subjects must present to Visit 6 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 6: Treatment 2 Follow-up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 6.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. | |
| 6.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. | |
| 6.3 | Compliance | Record the subject's compliance with wearing the study lenses. Note: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. | |
| 6.4 | PRO (CLUE and<br>MRD)<br>Questionnaires and<br>CLDEQ-8 | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO questionnaire. | |
| 6.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire | |
| 6.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. | 400 |
| 6.7 | Distance and Near<br>Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 6.8 | Visual Performance<br>Distance (4M)<br>Intermediate (64 cm)<br>Near (40 cm) | Visual performance will be recorded OD, OS, and OU for the following: Distance, Bright Illuminance High and Low Contrast ETDRS Charts 4M- HC#1, HC#2, HC#3 and LC#1, LC#2, | |

| | | LC#3 | |
|---|---|---|---|
| | | Near, Bright Illuminance Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast Near (40 cm) High Contrast and Low Contrast | |
| | | Distance, Dim Illuminance (with <u>Distance</u> goggles) High Contrast ETDRS Charts 4M-HC#4, HC#5, HC#6 Near, Dim Illuminance (with <u>Near</u> goggles) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near (40 cm). | |
| | | <ul> <li>Note:</li> <li>The room illuminance must be between 7.3 and 7.9 EV (394-597 lux).</li> <li>Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m2).</li> <li>Guillon-Poling, Near Chart Luminance Acceptable Range 10.8-11.1 EV (223-274 cd/m2).</li> <li>Do not use the Mesopic filter for Dim luminance (Dim luminance will be simulated by using the goggles)</li> </ul> | |
| 6.9 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix D |
| 6.10 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three | |

| - | iii | 294 22 76 | I |
|---|---|---|---|
| | | movement categories (primary gaze, upgaze, and push-up). | |
| | | If either lens is deemed unacceptable, the | |
| | | subject will be discontinued from the study. | |
| | | Remove the lenses, perform a slit-lamp | |
| | | evaluation, and complete the Final | |
| | | Evaluation form. | |
| 6.11 | Lens Deposits | Grade and record the amount of front and | |
| 6.10 | * *** 1.22. | back surface lens deposits for both eyes. | |
| 6.12 | Lens Wettability | Grade the wettability of the lens. | |
| 6.13 | Collection of | Collect unworn lenses returned by the | |
| | unworn lenses (if | subject. | |
| 6.14 | applicable) Lens Removal | II 411:4 4141-11 | |
| 0.14 | Lens Removal | Have the subject remove the study lenses and | |
| | | store in saline in a labeled glass vial. | |
| | | Note: The lenses do not need to be stored in | |
| | | a refrigerator. | |
| 6.15 | Biomicroscopy | Perform Biomicroscopy OD and OS. Slit | |
| 0.15 | Бюниеговеору | Lamp Classification Scales will be used to | |
| | | grade the findings. | |
| | | For the conjunctival redness 0.5 | A |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessmen | |
| | | will be graded in 1.0 increments. | |
| | | If any of these slit lamp findings are Grade 3 | |
| | | or higher, an AE must be recorded. All AEs | |
| | | must be followed to resolution. | |
| | | If the clearance of the fluorescein needs to be | |
| | | may be instilled. | |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. | |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Distance Subjective<br>Sphero-cylindrical<br>Refraction and<br>Distance Exit Visual<br>Acuity | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS, and OU). |
| F.2 | Subject Disposition | Indicate if the subject completed the study successfully. If subject discontinued from the study indicate the reason. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.
- Review of adverse event and concomitant medications.
- Documentation of any test article dispensed or collected from the subject, if applicable.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step Procedure Details | | |
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit |
| U.2 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. |
| U.3 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| U.4 | Entrance VA | Record the entrance distance and near visual acuity (OD, OS and OU). |

| Unscheduled Visit | | | |
|---|---|---|---|
| | | For near measures use the ETDRS 2000 | |
| | | Series Chart 1 or 2. | |
| | | The acuity will be recorded to the nearest | |
| | | letter OD, OS and OU. | - |
| U.5 | Subjective Sphero- | An optimal, binocular balanced distance | |
| | cylindrical Refraction | sphero-cylindrical refraction will be | |
| | | performed. | |
| | | Record the refraction and distance visual | |
| TIC | D' | acuity to the nearest letter. | |
| U.6 | Biomicroscopy | FDA Slit Lamp Classification Scale will be | |
| | | used to grade the findings | |
| | | For the conjunctival redness 0.5 | 5P 5% |
| | | unit increments will be used in the grading. | |
| | | Corneal Staining Assessment | |
| | | will be graded in 1.0 increments. | |
| | | If any of these slit lamp findings are Grade 3 | |
| | | or higher, an AE must be recorded. All AEs | |
| | | must be followed to resolution. | |
| | | States deligible from the control of the safe of the date of the control of the c | |
| | | If the clearance of the fluorescein needs to be | |
| | | expedited, preservative-free rewetting drops | |
| | | may be instilled. | |
| U.7 | Lens Dispensing | Additional study lenses may be dispensed | |
| 120319134 | S | when required. | |
| U.8 | Lens Fit Assessment: | Evaluate and grade lens centration, primary | |
| | | gaze movement, upgaze movement and | |
| | | tightness (push-up test). | |
| | | The subject should not proceed to wear the | |
| | | lenses if any of the following is observed: | |
| | | presence of limbal exposure (appearance) | |
| | | of clear cornea) in any gaze | |
| | | presence of edge lift | |
| | | presence of unacceptable movement | |
| | | (excessive or insufficient) in <u>all three</u> | |
| | | movement categories (primary gaze, | |
| | | upgaze, and push-up). | |
| | | If either lens is deemed unacceptable, the | |
| | | subject will be discontinued from the study. | |
| | | Remove the lenses, perform a slit-lamp | |

| | Unscheduled Visit | | |
|---|---|---|---|
| | | evaluation, and complete the Final Evaluation form. | 12.3 |
| U.9 | Exit Visual Acuity | Record the subject's exit distance and near visual acuity (OD, OS and OU). For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |

#### 7.4. Laboratory Procedures

Not Applicable

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

#### 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent
- they are eligible
- · completed all study visits

#### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject missed two consecutive study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study

- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the subject

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications and therapies are medications or therapies that contraindicate contact lens wear. See the Exclusion criteria for specific details.

#### 9.1. Systemic Medications

The following table lists the medications disallowed in this study.

Table 4: Disallowed systemic medications

| Class of Drug | Common Indication(s) | Common Examples |
|---|---|---|
| Anticholinergics | Irritable bowel syndrome, Parkinson's disease, peptic ulcer, cystitis, nasal congestion, cold symptoms, overactive bladder, COPD | Bentyl, Spiriva, Atrovent,<br>Hyosyne, Levsin, Symax Fastab,<br>Symax SL, Homax SL, Cogentin,<br>Transderm Scop, etc., |
| Oral<br>Phenothiazines | Antipsychotic disorders<br>(schizophrenia, mania) | Compazine, Mellarill, Thorazine, Phenagran, etc |
| Vitamin A<br>analogs | Cystic acne | Isotretinoin |
| Systemic/Topical<br>Corticosteroids | Arthritis, colitis, asthma,<br>bronchitis, allergic or<br>inflammatory conditions | Cortisone, Prednisone,<br>Hydrocortisone, Medrol, Kenalog<br>etc., |
| Oral Tetracycline | Urinary Tract Infection, acne,<br>chlamydia, gonorrhea | Sumcyin, Acitsite, Achromycin V, etc. |

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study then it must be reported to IEC/IRB. This is a "Major Deviation".

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature. The informed consent must also not be contradicted by the deviation.

Protocol waivers are prohibited

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

#### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Lens replacements that occur due to drops/fall-outs.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return (for test article return instructions).

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint

results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

**Serious Adverse Event (SAE)** – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Fetal distress, fetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater

- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other Grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation >2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

NOTE 1: to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

NOTE 2 to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

#### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment
  or study procedures and the adverse event (not related; unlikely related; possibly
  related; related see definition in Section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of
  intensity of the adverse event (mild; moderate; severe for all events see definition in
  Section 13.2.2).
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown.
- Actions Taken none; temporarily discontinued; permanently discontinued; other.

#### 13.2.1. Causality Assessment

Causality Assessment – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.
- Possibly Related An adverse event that might be due to the use of the test article, or
  to the study treatment or study procedures. An alternative explanation, e.g. concomitant
  treatment, concomitant disease(s), is inconclusive. The relationship in time is
  reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g.

concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

#### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

#### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements.

- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

#### 13.4.1. Reporting Adverse Events to Sponsor

#### **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All

subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

#### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

#### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

#### 13.4.3. Event of Special Interest

None
## 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

## 14. STATISTICAL METHODS

#### 14.1. General Considerations

All data summaries and statistical analyses will be performed using the SAS software version 9.4 (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (Descriptive statistics and/or frequency tables) will be provided by lens type for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

#### 14.2. Sample Size Justification

The study was powered to demonstrate non-inferiority of the Test lens relative to the Control with respect to binocular visual performance with minimum of 90% power and two-sided type I error of 5%. Assuming no difference between Test and Control, the required sample size to achieve non-inferiority for distance, intermediate and near visual performance at different lighting conditions are summarized in Table 5. The intra-class correlation (ICC) and standard deviations (STD) used in the sample size calculations were from a similar study (CR6267). The sample size calculations were conducted using the SAS procedure PROC POWER for paired t-test.

Table 5: Required sample to achieve non-inferiority

| Distance | Lighting Condition | STD<br>Test | STD<br>Control | ICC | Sample<br>Size |
|---|---|---|---|---|---|
| Distance | High Luminance High Contrast | 0.091 | 0.094 | 0.60 | 31 |
| | High Luminance Low Contrast | 0.091 | 0.105 | 0.68 | 29 |
| | Low Luminance High Contrast with Distance Goggles | 0.101 | 0.092 | 0.64 | 31 |

| Intermediate | High Luminance High Contrast | 0.095 | 0.116 | 0.68 | 34 |
|---|---|---|---|---|---|
| | High Luminance Low Contrast | 0.107 | 0.129 | 0.71 | 38 |
| | Low Luminance High Contrast with Near Goggles | 0.125 | 0.152 | 0.81 | 36 |
| Near | High Luminance High Contrast | 0.086 | 0.113 | 0.63 | 36 |
| | High Luminance Low Contrast | 0.103 | 0.130 | 0.69 | 40 |
| | Low Luminance High Contrast with Near Goggles | 0.115 | 0.137 | 0.73 | 40 |

STD: standard deviation, ICC: intra-class correlation

After adjusting for 7% drop-outs or lost to follow-up, the plan is to enroll 48 subjects with a target completion of 40 subjects.

# 14.3. Analysis Populations

The following analysis populations will be defined and used in the analysis and presentation of the data.

#### All Enrolled:

All Enrolled Population includes all subjects with recorded data in the electronic Case Report Form (eCRF) database

# **Intent-To-Treat (ITT):**

Intent-to-treat will include all the subjects who were randomized to study treatment. Subjects will be analyzed as per randomized treatment. At least one observation should be recorded. Discontinued subjects, subjects with major protocol deviations and ineligible subjects who were inadvertently randomized will be included in the ITT analyses.

# **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation for safety endpoints should be recorded (e.g. ocular symptom, slit-lamp finding, etc.) or on after treatment start date. Subjects will be analyzed as per treatment received.

#### Per Protocol (PP)

All subjects who have successfully completed the study and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock. Justification of excluding subjects with protocol deviations from the per-protocol population set will be documented in a memo to file.

The primary analysis will be conducted on the per-protocol population. A sensitivity analysis will be conducted on the ITT population.

# 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

## 14.5. Primary Analysis

## Visual Performance:

Binocular visual performance at 2-week follow-up visit will be analyzed separately by lighting condition and distance using a Bayesian repeated measurement random-effects model to compare between Test and Control lenses. Each regression model will include baseline values, lens type, lens wearing sequence and lens wearing period as fixed effects and investigational site as random effect. Other subject characteristics such as age, gender will be included as fixed effects when appropriate. Unstructured covariance matrix will be used to model the residual errors among observations within subjects. Non informative prior distributions will be used for the coefficients in the models as well as for the error terms. Independent vague normal N(0,1000) priors will be used for the regression coefficients, inverse gamma IG(0.001, 0.001) for the variance of the random effect site and inverse Wishart for the residual errors. A Markov-Chain Monte Carlo (MCMC) sampling algorithm will be used to carry out the marginal posterior distributions of the parameters. Results will be reported as regression coefficient mean estimates with 95% credible intervals.

The null and alternative hypotheses for non-inferiority of Test lens relative to Control are as follows:

*H*0:  $\Delta > 0.05$  *HA*:  $\Delta < 0.05$ 

where  $\Delta$  is the posterior mean difference in visual performance between Test and Control (Test minus Control). Non-inferiority will be declared if the upper bound of the credible interval of the posterior mean difference is less than 0.05.

The primary analysis will be conducted on the per-protocol population. A sensitivity analysis will be conducted on the ITT population.

#### 14.6. Secondary Analysis

All secondary endpoints will be summarized with descriptive statistics at baseline and followup visits for each study lens type. Safety variables will be summarized on safety population and efficacy variables on both per-protocol and ITT populations.

#### 14.7. Other Exploratory Analyses

## Comfort and Vision CLUE Scores

CLUE comfort and vision CLUE scores will be analyzed separately using the same statistical method described in the primary analysis. Posterior mean differences ( $\delta$ ) in CLUE scores between Test and Control will be calculated with 95% credible intervals. The probability of achieving non-inferiority using a margin of -5 point in the CLUE scale,  $Pr(\delta \ge -5 \mid data)$ , will be calculated.

Further exploratory analysis will be conducted if necessary, at the discretion of the Study Responsible Clinician.

# 14.8. Interim Analysis

No interim analysis is planned in this study

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis may be conducted using multiple imputation methods. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 20 imputations.

# 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

## 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

## 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External Data Sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual

Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

# 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 15 15.3 ClinicalTrials.gov

This trial will be registered on clincaltrials.gov

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

## 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The

Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

# 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

### 18. ETHICAL AND REGULATORY ASPECTS

# 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

# 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

# 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

# 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>5</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps

should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

# 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- 6. EU MDR 2017/745
- 7. Wirth, R.J., et al., Development of the Contact Lens User Experience: CLUE Scales. Optom Vis Sci, 2016. 93(8): p. 801-8.

APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)












# Clinical Study Protocol Johnson & Johnson Vision Care, Inc.

APPENDIX B: PATIENT INSTRUCTION GUIDE (TO BE PROVIDED SEPARATELY)

IMPORTANT: Please read carefully and keep this information for future use.

This Package Insert and Fitting Instruction Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



1-DAY ACUVUE® MOIST Brand Contact Lenses 1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM 1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses

> etafilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily Disposable Wear



CAUTION: U.S. Federal law restricts this device to ROnly CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner.

CR-6372, v 2.0


# SYMBOLS KEY

The following symbols may appear on the label or packaging:

| SYMBOL | DEFINITION |
|--------------|-----------------------------------------------------|
| Ţ <u>i</u> | Consult Instructions for Use |
| ••• | Manufacturer |
| س | Date of Manufacture |
| $\square$ | Use By Date (expiration date) |
| LOT | Batch Code |
| STERILE | Sterilized Using Steam Heat |
| 8 | Do Not Re-Use (Single Use) |
| ₩ <b>(</b> ) | Lens Orientation Correct |
| ₩ X | Lens Orientation Incorrect (Lens Inside Out) |
| C€<br>0086 | Quality System Certification Symbol |
| 0 | Fee Paid for Waste Management |
| EC REP | Authorized Representative in the European Community |

Visit www.acuvue.com/guides for additional information about symbols.

# DESCRIPTION

1-DAY ACUVUE® MOIST Brand Contact Lenses, 1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM, and 1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are soft (hydrophilic) contact lenses available as spherical, toric, or multifocal lenses, and include LACREON® Technology.

The lens material (etaflicon A) is a copolymer of 2-hydroxyethyl methacrylate and methacrylic acid cross-linked with 1, 1, 1-trimethylol propane trimethacrylate and ethylene glycol dimethacrylate.

2

CR-6372, v 2.0


The lenses are tinted blue using Reactive Blue Dye #4 to make the lenses more visible for handling. A benzotriazole UV absorbing monomer is used to block UV radiation.

#### Lens Properties:

The physical/optical properties of the lens are:

 Specific Gravity (calculated): 0.98 – 1.12 1.40 Refractive Index: Light Transmittance: 85% minimum Surface Character: Hydrophilic Water Content: 58%

Oxygen Permeability (D/k):

METHOD VALUE

21.4 x 10 <sup>11</sup> (cm²/sec) (ml O<sub>2</sub>/ml x mm Hg) @ 35°C Fatt (boundary corrected, edge corrected)

28.0 x 10 11 (cm<sup>2</sup>/sec) Fatt (boundary corrected, non-edge corrected)

(ml O<sub>2</sub>/ml x mm Hg) @ 35°C

### Lens Parameters Ranges:

 Diameter (DIA): 12.0 mm to 15.0 mm Varies with power Center Thickness: • Base Curve (BC): 7.85 mm to 10.00 mm
• Spherical Power (D): -20.00D to +20.00D Cylinder Power (CYL): -0.25D to -10.00D 2.5° to 180° Axis (AXIS): ADD Powers: +0.25D to +4.00D

# **AVAILABLE LENS PARAMETERS**

1-DAY ACUVUE® MOIST Brand Contact Lenses are hemispherical shells of the following dimensions:

Diameter (DIA): 14.2 mm

Center Thickness: 0.084 mm to 0.230 mm (varies with power)

3

CR-6372, v 2.0


Base Curve (BC): 8.5 mm, 9.0 mm

-0.50D to -6.00D (in 0.25D increments) -6.50D to -12.00D (in 0.50D increments) Powers (D):

+0.50D to +6.00D (in 0.25D increments)

1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM are hemitoric shells of the following dimensions:

Diameter (DIA): 14.5 mm

Center Thickness: 0.090 mm to 0.189 mm (varies with power)

Base Curve (BC): 8.5 mm

+0.00 to -6.00D (in 0.25D increments) Powers (D):

Cylinders (CYL): -0.75D, -1.25D, -1.75D, -2.25D\* Axis (AXIS): 10° to 180° in 10° increments \*-2.25D cylinder is available in 10°, 20°, 70°, 80°, 90°,

100°, 110°, 160°, 170°, 180° axes only

-6.50D to -9.00D (in 0.50D increments)

Cylinders (CYL): -0.75D, -1.25D, -1.75D, -2.25D\* Axis (AXIS): 10°, 20°, 60°, 70°, 80°, 90°, 100°, 110°, 120°, 160°, 170°, 180°

 $^*\mbox{-}2.25\mbox{D}$  cylinder is available in 20°, 90°, 160°, 180°

axes only

+0.25D to +4.00D (in 0.25D increments) Cylinders (CYL): -0.75D, -1.25D, -1.75D

Axis (AXIS): 10°, 20°, 70°, 80°, 90°, 100°, 110°, 160°,

170°, 180°

1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are hemispherical shells of the following dimensions:

Center Thickness: 0.084 mm to 0.207 mm (varies with power)

Base Curve (BC): 8.4 mm

Powers (D): +6.00D to -9.00D (in 0.25D increments) Near ADD Powers Low Near ADD (LOW): +1.25D (MAX ADD): Medium Near ADD (MID): +1.75D

High Near ADD (HGH): +2.50D

4

CR-6372, v 2.0


# TRANSMITTANCE CURVES

1-DAY ACUVUE $^{9}$  MOIST Brand Contact Lenses (etaflicon A) Visibility Tinted with UV Blocker vs. 24 yr. old human cornea and 25 yr. old human crystalline lens.



 $^*$ The data are representative measurements taken through the central 3-5 mm portion for the thinnest marketed lens (-3.00D lens, 0.084 mm center thickness).

 Lerman, S., Radiant Energy and the Eye, MacMillan, New York, 1980, p. 58, figure 2-21
 Waxler, M., Hitchins, V.M., Optical Radiation and Visual Heath, CRC Press, Boca Raton, Florida, 1986, p. 19, figure 5

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

### **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays on the retina.

The UV Blocking for these lenses averages 97% in the UVB range of 280 nm to 315 nm and 82% in the UVA range of 316 nm to 380 nm for the entire power range.

5

CR-6372, v 2.0


NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

# **INDICATIONS (USES)**

1-DAY ACUVUE® MOIST Brand Contact Lenses are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 1.00D or less of astiomatism.

1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 0.50D to 3.00D of astigmatism.

1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are indicated for daily disposable wear for the optical correction of distance and near vision in presbyopic phakic or aphakic persons with non-diseased eyes who may have 4.00D of ADD power or less and 0.75D or less of astigmatism.

The lenses contain a UV Blocker to help protect against transmission of harmful UV radiation to the cornea and into the eye.

When prescribed for daily disposable use, no cleaning or disinfection is required. Lenses should be discarded upon removal.

# CONTRAINDICATIONS (REASONS NOT TO USE)

DO NOT USE these lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the eye
- Any eye disease, injury, or abnormality that affects the cornea, conjunctiva, or eyelids.
- · Severe insufficiency of lacrimal secretion (dry eye).
- Corneal hypoesthesia (reduced corneal sensitivity).

6

CR-6372, v 2.0


- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
- Ocular irritation due to allergic reactions which may be caused by use
  of contact lens solutions (i.e., rewetting drops) that contain chemicals or
  preservatives (such as mercury, Thimerosal, etc.) to which some people
  may develop an allergic response.
- Any active corneal infection (bacterial, fungal, protozoal, or viral).
- If eyes become red or irritated.

### **WARNINGS**

Patients should be advised of the following warnings pertaining to

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION. IF THE PATIENT EXPERIENCES:

- · Eye Discomfort,
- Excessive Tearing,
- · Vision Changes,
- . Loss of Vision,
- · Eye Redness, or
- . Other Eye Problems,

THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

- When prescribed for daily wear, patients should be instructed not to wear their lenses while sleeping. Clinical studies have shown that when lenses are worn overnight, the risk of ulcerative keratitis is greater than among those who do not wear them overnight.<sup>3</sup>
- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products are essential for the safe use of these products.

7

CR-6372, v 2.0


 The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care.

<sup>3</sup>New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

### Specific Instructions for Use and Warnings:

# Water Activity

### Instruction for Use

Do not expose contact lenses to water while wearing them.

#### WARNING:

Water can harbor microorganisms that can lead to severe infection, vision loss, or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving

# **PRECAUTIONS**

### Special Precautions for Eye Care Professionals:

 Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers.
 Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.

 Patients who wear these lenses to correct presbyopia using monovision (or modified monovision using 1-DAY ACUVUE® MOIST Brand MULTIFOCAL) may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.

8

CR-6372, v 2.0


- Fluorescein, a yellow dye, should not be used while the lenses are on the eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used in eyes, the eyes should be flushed with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove lenses immediately if the eyes become red or irritated.

Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions.

### **Handling Precautions:**

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps, creams, deodorants, or sprays in the eyes or on the lenses. It is best to put on lenses before putting on makeup.
- DO NOT touch contact lenses with the fingers or hands if the hands are not free of foreign materials, as microscopic scratches of the lenses may occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the Patient instruction Guide for these lenses and those prescribed by the Eye Care Professional.
- · Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens container. Slide the lens up the side of the bowl until it is free of the container.
- Do not touch the lens with fingernails.

### **Lens Wearing Precautions:**

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for Sticking (Non-Moving) Lenses." The lens should move freely on the eye for the continued health of the eye. If nonmovement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional

9

CR-6372, v 2.0


- The patient should be advised to never allow anyone else to wear their lenses. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hairspray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- Avoid all harmful or irritating vapors and fumes while wearing lenses.

### Lens Care Precautions:

 The patient should be informed that no cleaning or disinfection is needed when lenses are worn for daily disposable wear. Patients should always dispose of lenses when removed and have spare lenses or spectacles available.

### Other Topics to Discuss with Patients:

- Always contact the Eye Care Professional before using any medicine in the eyes
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- As with any contact lens, follow-up visits are necessary to assure the continuing health of the patient's eyes. The patient should be instructed as to a recommended follow-up schedule.

### Who Should Know That the Patient is Wearing Contact Lenses?

- Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.
- Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

10

CR-6372, v 2.0


# ADVERSE REACTIONS

The patient should be informed that the following problems may occur when wearing contact lenses:

- The eye may burn, sting, and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ulcers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis, and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eve.
- Poor visual acuity, blurred vision, rainbows or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:

- How do the lenses feel on my eyes?
- · How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be advised that when any of the above symptoms occur, a serious condition such as infection, corneal ulcer, neovascularization, or iritis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eve damage.

11

CR-6372, v 2.0


# **GENERAL FITTING GUIDELINES**

### A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- · Motivation to wear lenses
- Ability to follow instructions regarding lens wear
- General health
- · Ability to adequately handle and care for the lenses
- · Ability to understand the risks and benefits of lens wear

Patients who do not meet the above criteria should not be provided with contact lenses.

### B. Pre-fitting Examination

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), keratometry, and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the lens fitting instructions as outlined below.

#### C. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than  $\pm 4.00D$ .

### D. Base Curve Selection (Trial Lens Fitting)

The following trial lenses should be selected for patients regardless of keratometry readings. However, corneal curvature measurements should be performed to establish the patient's baseline ocular status.

12

CR-6372, v 2.0


- 1-DAY ACUVUE® MOIST: 8.5 mm/14.2 mm
- 1-DAY ACUVUE® MOIST for ASTIGMATISM: 8.5 mm/14.5 mm
- 1-DAY ACUVUE® MOIST MULTIFOCAL: 8.4 mm/14.3 mm

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

### 1. Criteria of a Properly Fit Lens

A properly fit lens will center and completely cover the cornea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

### 2. Criteria of a Flat Fitting Lens

A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete corneal coverage (i.e., limbal exposure), excessive movement with the blink and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

### 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with the lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

### E. Final Lens Power (Spherical)

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct lens power unless there is excessive residual astigmatism.

13

CR-6372, v 2.0


| Example 1 | |
|----------------------------|------------------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |
| Example 2 | |
| Example 2 | |
| Example 2 Diagnostic lens: | -2.00D |
| • | -2.00D<br>+0.25D |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see **PATIENT MANAGEMENT** section).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

# TORIC FITTING GUIDELINES

Although most aspects of the fitting procedure are identical for all types of soft contact lenses, including toric lenses, there are some additional steps and/or rules to follow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing 1-DAY ACUVUE® MOIST for ASTIGMATISM are that you must determine the stability, repeatability, and drift angle of the lens axis so that you can prescribe the correct lens axis for the patient.

### A. How to Determine Lens Cylinder and Axis Orientation

#### 1. Locate the Orientation Marks

To help determine the proper orientation of the toric lens, you'll find two primary marks approximately 1 mm from the lens edge representing the vertical position on opposite ends of the lens at 6 and 12 o'clock (Fig. 1). Because of the lens' ballasting system, either mark can represent the vertical position – there is no "top" and "bottom" as in a prism-ballasted lens. You don't need to view both marks to assess orientation; simply look for the 6 o'clock mark as you would with a prism-ballasted lens.

14

CR-6372, v 2.0




You'll need a slit lamp biomicroscope with a 1 to 2 mm parallelepiped beam to highlight the marks when the lens is fitted to the eye. There are a number of techniques you can use to improve the visibility of the 6 o'clock mark. Using a parallelepiped beam and medium magnification (10x or 15x), slowly pan down the lens, looking just below the direct illumination at the retroilluminated area. Backlighting the mark this way should make it more visible. Sometimes manipulating the lower lid may be necessary to uncover the mark.

### 2. Observe Lens Rotation and Stability

Observe the position and stability of the "bottom" mark. It usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable.

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still enable you to fit a toric lens for that eye, as long as the lens always returns to the same "drift axis" position after settling. The deviation can be compensated for in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 o'clock, this position must be stable and repeatable. With full eye movement or heavy blink, you may see the marks swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

### 3. Assessing Rotation

Imagine the eye as a clock dial and every hour represents a 30° interval. If the orientation mark of the initial lens stabilizes somewhat left or right of the vertical position, the final lens will orient on the eye with the same deviation. You can use an axis reticule in the slit lamp or use a line-scribed lens in a spectacle trial frame to measure or estimate the "drift angle" of the cylinder axis.

To compensate for this "drift," measure or estimate the "drift," then add or subtract it from the refractive axis to determine the correct cylinder axis. Use the LARS (Left Add, Right Subtract) method to determine which direction to compensate.

15

CR-6372, v 2.0


#### **B. Final Lens Power**

When the diagnostic lens has its axis aligned in the same meridian as the patient's refractive axis, a spherocylindrical over-refraction may be performed and visual acuity determined. However, in the case of crossed axes, such as when the diagnostic lens axis is different from the spectacle cylinder axis, it is not advisable to perform a full spherocylindrical over-refraction because of the difficulty in computing the resultant power. A spherical over-refraction without cylinder refraction may be performed.

If the required cylinder correction falls between two available cylinder powers, it is recommended to prescribe the lower cylinder power lens. See below for instructions on how to determine the final lens power.

### 1. For the Sphere

If sphere alone or combined sphere and cylinder Rx > 4.00D, compensate for vertex distance. If sphere alone or combined sphere and cylinder Rx  $\leq$   $\pm$ 4.00D, vertex compensation is not necessary.

#### 2. For the Cylinder

Adjust the axis by the drift angle using the LARS method. Choose a cylinder that is  $\leq 0.50D$  from the refractive cylinder.

### 3. Case Examples

### Example 1

Manifest (spectacle) refraction:

O.D. -2.50D / -1.25D x 180° 20/20

O.S. -2.00D / -1.00D x 180° 20/20

Choose a diagnostic lens for each eye with axis 180°. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'clock position on both eyes, choose the appropriate cylinder as listed previously. If the lens has not yet stabilized, recheck until stable.

Here is the Rx prescribed:

O.D. -2.50D / -1.25D x 180°

O.S. -2.00D / -0.75D x 180°

16

CR-6372, v 2.0


#### Example 2

Manifest (spectacle) refraction: O.D. -3.00D / -1.00D x 90° 20/20 O.S. -4.75D / -2.00D x 90° 20/20

Choose diagnostic lenses of -3.00D / -0.75D x 90° for the right eye and -4.50D / -1.75D x 90° for the left eye, the nearest lenses available to the spherical power and axis needed. For the left eye, since the manifest refraction called for -4.75D, compensating for vertex distance the sphere is reduced by 0.25D to -4.50D. The cylinder power will be -1.75D. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

### Right Eve

The orientation mark on the right lens rotates left from the 6 o'clock position by  $10^\circ$  and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate the 10° axis drift by adding it to the manifest refraction axis.

Here is the Rx prescribed: O.D. -3.00D / -0.75D x 100°

#### Loff Evo

The orientation mark on the left lens rotates right from the 6 o'clock position by 10° and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate for the  $10^{\circ}$  axis drift by subtracting it from the manifest refraction axis.

Here is the Rx prescribed: O.S. -4.50D / -1.75D x 80°

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see PATIENT MANAGEMENT section).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

17

CR-6372, v 2.0


### MULTIFOCAL FITTING GUIDELINES

### A. Presbyopic Needs Assessment & Patient Education

Multifocal contact lenses may produce compromise to vision under certain circumstances and the patient should understand that they might not find their vision acceptable in specific situations (i.e., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments. Occupational and environmental visual demands should be considered. If the patient requires critical visual acuity and stereopsis, it should be determined by trial whether this patient can function adequately with 1-DAY ACUVUE® MOIST MULTIFOCAL. Wearing these lenses may not be optimal for activities such as:

- Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- Driving automobiles (e.g., driving at night). Patients who cannot meet
  their state driver's license requirements with the 1-DAY ACUVUE® MOIST
  MULTIFOCAL should be advised to not drive with this correction, OR may
  require that additional over-correction be prescribed.

1-DAY ACUVUE® MOIST MULTIFOCAL is not recommended for patients who have -1.00D or greater of refractive cylinder as this level of uncorrected cylinder may lead to additional visual compromise. These lenses are available in the following ADD powers:

- Lens "LOW" = low near ADD lens (Max ADD +1.25)
- Lens "MID" = medium near ADD lens (Max ADD +1.75)
- Lens "HGH" = high near ADD lens (Max ADD +2.50)

#### **B. Initial Power Determination**

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than ±4.00D. Determine the spherical equivalent distance prescription for a multifocal patient. Determine the eye dominance using one of the methods below:

18

CR-6372, v 2.0


Method 1 Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

Method 2 Determine which eye does not accept added plus power. Place a +1.00D hand-held trial lens in front of one eye and then the other while the distance refractive error correction is in place for both eyes while the patient is viewing the distance visual acuity chart. The eye with the plus over it that the patient notices the greatest reduction in vision is determined to be the dominant eye.

### C. Select the Initial Trial Lens

- For each eye, select the trial lens distance power that is closest to the
  patient's distance spherical equivalent. Remember to compensate for
  vertex distance if the refraction is greater than ±4.00D.
- Select the near power of the lens based on the patients ADD range as follows:
  - ADD: +0.75D to +1.25D use a low near ADD (LOW) lens on each eye
  - ADD: +1.50D to +1.75D use a medium near ADD (MID) lens on each eye
  - ADD: +2.00D to +2.50D use a medium near ADD (MID) on the dominant eye and a high near ADD (HGH) lens on the non-dominant eye
- 3. Allow the lenses to settle for a minimum of 10 minutes.
- 4. Assess distance and near vision binocularly and monocularly.
- Demonstrate the vision under various lighting conditions (normal and decreased illumination) and at distance, intermediate, and near.
- Make adjustments in power as necessary based on the distance overrefraction. The use of hand-held trial lenses is recommended. Check the impact on distance and near vision.
- 7. If vision is still unacceptable, make adjustments in power as necessary (see "Multifocal Troubleshooting" below). If distance and near vision are acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see PATIENT MANAGEMENT section).

19

CR-6372, v 2.0


#### D. Multifocal Troubleshooting

#### **Unacceptable Near Vision**

If it has been determined that no change is required based on the overrefraction, then add +0.25D to the spherical power of the non-dominant eye.

### **Unacceptable Distance Vision**

If it has been determined that no change is required based on the overrefraction, then make the changes as listed below:

- If the patient is wearing two "LOW" ADD lenses, change the dominant eye to a 1-DAY ACUVUE® MOIST sphere lens with a power equal to the spherical equivalent distance prescription.
- If the patient is wearing two "MID" ADD lenses, change the ADD power in the dominant eye to the "LOW" ADD power.
- If the patient is wearing a "MID" ADD lens in the dominant eye and a "HGH" ADD lens in the non-dominant eye, change the non-dominant eye to a "MID" ADD lens and add +0.25D to the distance power.

#### E. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches and a feeling of slight imbelance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

20

CR-6372, v 2.0


# MONOVISION FITTING GUIDELINES

#### A. Patient Selection

### 1. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

- Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- Driving automobiles (e.g., driving at night). Patients who cannot meet
  their state driver's license requirements with monovision correction
  should be advised to not drive with this correction, OR may require that
  additional over-correction be prescribed.

#### 2. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g., reading a menu in a dimly lit restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision, and straight ahead and upward gaze that monovision contact lenses provide.

21

CR-6372, v 2.0


#### B. Eye Selection

### 1. Ocular Preference Determination Methods

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

Method 1 Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

Method 2 Determine which eye will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eve and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

### 2. Other Eye Selection Methods

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

### Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

### Visual Demands Method

Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example: A secretary who places copy to the left side of the desk will function best with the near lens on the left eye.

#### C. Special Fitting Characteristics

### 1. Unilateral Vision Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens, whereas a bilateral myope would require corrective lenses on both eyes.

22

CR-6372, v 2.0


#### Examples

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left eye uncorrected for near.

### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

#### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the **GENERAL FITTING GUIDELINES** for base curve selection described in this Packane Insert

Case history and a standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next, determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernalis. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed, should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

23

CR-6372, v 2.0


An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

### D. Other Suggestions

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Have supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet state driver's licensing requirements with monovision correction.
- Make use of proper illumination when carrying out visual tasks.

24

CR-6372, v 2.0


Monovision fitting success can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of clear near vision, and straight ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

# PATIENT MANAGEMENT

- Follow the accepted standard of care in fitting and following up with your patient, e.g., American Optometric Association standard of care.
- Schedule the appropriate follow-up examination.
- Preferably, at the follow-up visits, lenses should have been worn for at least six hours.
- Provide the patient with a copy of the PATIENT INSTRUCTION GUIDE for these lenses, which can be found at www.acuvue.com. REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULES.

# WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to over wear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.

25

CR-6372, v 2.0


The maximum suggested wearing time for these lenses is:

| DAY | HOURS |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

# REPLACEMENT SCHEDULE

These lenses are indicated for daily disposable wear and should be discarded upon removal.

When disposed of after a single daily use, these lenses may reduce the risk of developing giant papillary conjunctivitis.  $^4$ 

When worn as a daily disposable lens, these lenses may provide improved comfort for many patients who experience mild discomfort and itching associated with allergies during contact lens wear, compared to lenses replaced at intervals of greater than 2 weeks.

Clinical research has shown that when worn on a daily disposable basis, these lenses may provide improved comfort for 2 out of 3 patients who reported suffering from discomfort associated with allergies during contact lens wear.

# LENS CARE DIRECTIONS

The Eye Care Professional should review with patients that no cleaning or disinfection is needed with daily disposable lenses. Patients should always dispose of lenses when they are removed and have replacement lenses or spectacles available.

For complete information concerning contact lens handling and care, refer to the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

### Care for Sticking (Non-Moving) Lenses

During removal, if the lens sticks to the eye, the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution

2

CR-6372, v 2.0


<sup>&</sup>lt;sup>4</sup>The CLAO Journal, July 1999, Volume 25, Number 3

directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should **immediately** consult the Eye Care Professional.

### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

### **HOW SUPPLIED**

Each UV-absorbing sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with povidone. The plastic package is marked with the following:

- 1-DAY ACUVUE® MOIST: base curve, power, diameter, lot number, and expiration date
- 1-DAY ACUVUE® MOIST for ASTIGMATISM: base curve, power, diameter, cylinder, axis, lot number, and expiration date
- 1-DAY ACUVUE® MOIST MULTIFOCAL: base curve, power, diameter, ADD power, lot number, and expiration date

# REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with these lenses should be reported to:

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acuvue.com

27

CR-6372, v 2.0


Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-600-843-2020 www.acuvue.com



©Johnson & Johnson Vision Care, Inc. 2017 In Canada: Johnson & Johnson Vision Care division of Johnson & Johnson Inc. In USA: Johnson & Johnson Vision Care, Inc. Printed in USA Revision date: 07/17 Revision number: M-07-17-02

1-DAY ACUVUE® MOIST and LACREON® are Trademarks of Johnson & Johnson Vision Care, Inc.

CR-6372, v 2.0


APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

#### APPENDIX D: BINOCULAR OVER REFRACTION



#### APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE



#### APPENDIX F: OCULAR DOMINANCE



#### APPENDIX G: LENS FITTING GUIDE

| F |
|---|



### APPENDIX H:

- LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS
- EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING
- DETERMINATION OF NEAR ADD
- NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE
- LENS FITTING CHARACTERISTICS
- SUBJECT REPORTED OCULAR SYMPTOMS
- FRONT AND BACK SURFACE LENS DEPOSIT GRADING
  PROCEDURE
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL
  REFRACTIONS
- BIOMICROSCOPY SCALE
- KERATOMETRY
- DISTANCE AND NEAR VISUAL ACUITY EVALUATION
- ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE
- PATIENT REPORTED OUTCOMES
- WHITE LIGHT LENS SURFACE WETTABILITY
- VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS










**Attachment A** Efron Grading Scale for Limbal Redness (0.5 unit increments)



Attachment B Efron Grading Scale for Limbal Redness (1.0 unit increments)








#### Attachment E




#### EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING









#### **DETERMINATION OF NEAR ADDITION**



























NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE






#### LENS FITTING CHARACTERISTICS





CR-6372, v 2.0






Attachment B Example of Evaluation of Primary Gaze Movement





## SUBJECT REPORTED OCULAR SYMPTOMS/PROBLEMS



FRONT AND BACK SURFACE LENS DEPOSIT GRADING PROCEDURE



CR-6372, v 2.0



### Attachment A



### Attachment B




### Attachment C



DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS












CR-6372, v 2.0











CR-6372, v 2.0






CR-6372, v 2.0






CR-6372, v 2.0




CR-6372, v 2.0




KERATOMETRY PROCEDURE



## DISTANCE AND NEAR VISUAL ACUITY EVALUATION








DISTANCE LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE









### WHITE LIGHT LENS SURFACE WETTABILITY





VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION






### APPENDIX A: CHART LUMINANCE VERIFICATION LOG



### APPENDIX C: CONVERSION TABLE FOR "EV' TO "LUX" FOR ROOM ILLUMINATION



### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6372 Clinical Evaluation of a Reusable Multifocal Optical Design in a Presbyopic Population Phase II

Version and Date: 2.0 25 October 2019

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |

CR-6372, v 2.0 JJVC CONFIDENTIAL